CLINICAL TRIAL: NCT00351000
Title: An Open Label Trial of Ziprasidone as an Adjuvant for Clozapine- or Olanzapine-Associated Diabetes Mellitus or Impaired Fasting Glucose in Chronic Schizophrenia
Brief Title: Ziprasidone for Clozapine- or Olanzapine-Associated Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Suffolk Mental Health Association (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, David C. Henderson, MD, Associate Professor of Psychiatry, Harvard Medical School (HMS and HSDM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-2005
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Ziprasidone; Diabetes; Insulin Resistance
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus; Insulin Resistance | interventions — ziprasidone

INTERVENTIONS:
Drug: Ziprasidone

SUMMARY:
This study is a six-week, open label trial of the novel antipsychotic agent, ziprasidone, added to a stable dose of clozapine or olanzapine in 40 diabetes mellitus patients, patients with an impaired fasting glucose or insulin resistance with schizophrenia or schizoaffective disorder. The first two weeks will be a fixed-dose of ziprasidone 40 mg twice a day. During weeks 2-6, the ziprasidone dose may be increased up to 80 mg twice a day.

DETAILED DESCRIPTION:
Specific Aims:

This study is a six-week, open label trial of the novel antipsychotic agent, ziprasidone, added to a stable dose of clozapine or olanzapine in 40 diabetes mellitus patients, patients with an impaired fasting glucose or insulin resistance with schizophrenia or schizoaffective disorder.

STUDY PROCEDURES:

We have designed this trial to examine effects upon weight, lipids and glucose metabolism along with positive symptoms, negative symptoms, and depressive symptoms during a six-week open label study.

Location:

This study will be performed at the Freedom Trail Clinic by faculty of the Schizophrenia Program of the Massachusetts General Hospital and staff of the Freedom Trail Clinic.

Subjects:

Subjects will include 40 outpatients with schizophrenia or schizoaffective disorder treated with clozapine or olanzapine for at least one year. Twenty clozapine-treated subjects and twenty olanzapine-treated subjects with type 2 diabetes mellitus, impaired fasting glucose, or insulin resistance will be recruited. Patients will be excluded for significant medical illness, seizure disorder, substance abuse, or inability to provide informed consent.

Methods:

Medication Trial:

Patients will be treated with open label ziprasidone 40 mg 2x/day for the first 2 weeks. After 2 weeks the study drug may be increased up to ziprasidone 80 mg 2x/day. The clozapine or olanzapine dose will be unchanged during the trial. Patients will be given a two-week supply of medication at baseline and weeks 2 and 4 with additional capsules for study drug compliance and accountability. Following completion of the trial patients will have the option of continuing the ziprasidone. Subjects will return 4 weeks following study completion to examine whether any observed changes are persistent. Additionally, patients will be assessed at a 3 month follow-up post their 10 week assessment for metabolic changes.

Screening Visit The diagnosis of schizophrenia or schizoaffective disorder will be confirmed by a research psychiatrist using DSM IV criteria. A physical examination will be performed and medical history, vital signs, weight, waist/hip circumference, EKG and demographic information will be obtained. Demographic information will also include the date of onset or the duration of diabetes mellitus. Laboratory measures will include a CBC, fasting glucose, insulin, cholesterol (total, HDL and LDL), triglycerides, hemoglobin A1C and leptin. Plasma will also be obtained for assay of clozapine, norclozapine, or olanzapine concentrations at the screening visit.

Baseline Assessment:

The following scales will be completed at baseline and will comprise the treatment efficacy battery: Positive and Negative Syndrome Scale (PANSS), Scale for Assessment of Negative Symptoms (SANS), Clinical Global Impression Scale (CGI), Hamilton Depression Rating Scale (HAM-D), Global Assessment Scale (GAS), Fatigue Scale Inventory (FSI) and the Quality of Life Scale (QOL).

Safety Assessments:

Vital signs, weight, and waist/hip circumference will be performed at each visit (weeks 0, 2, 4, 6 and 10 and at the 3 month follow-up). Side effects will be monitored at baseline and weeks 2, 4, 6 and 10 using the SAFTEE (Levine and Schooler 1986). EPS will be evaluated at baseline and weeks 2, 4, 6 and 4 week follow-up using the Simpson-Angus Scale, Barnes Akathisia Scale, and the Abnormal Involuntary Movement Scale (AIMS). EKG will be performed at baseline, weeks 2, 4, 6, and 10. A patient will be discontinued from the study if their QTc interval is greater than 450. Changes in medication will be recorded throughout the study including changes to diabetes medication (weeks 0, 2, 4, 6 and 10 and at the 3-month follow-up).

Energy Expenditure and Dietary Assessment:

Patients will be asked to wear an accelerometer (Actigraph model 7164) to obtain an objective measure of physical activity. This is single channel accelerometer which measures and records vertical accelerations ranging from 0.05 to 2 G's with a frequency response of 0.25 to 2.50 hertz. These parameters detect normal body motion and filter out high frequency movement such as vibrations. The accelerometer is positioned at the waist and worn for four consecutive days except during sleep or while in water (i.e. swimming or taking a shower). The raw data is then read and processed by a custom data processing program to estimate energy expenditure. Patients will be instructed to complete a four-day food record to assess dietary intake. Food records will be reviewed for completeness and analyzed using Nutrition Data System (NDS). Energy expenditure and dietary intake will be assessed at baseline, weeks 4 and 6 and at the 3 month follow-up.

Subject Recruitment:

The Freedom Trail Clinic has well established procedures for identifying, referring and recruiting subjects for research. Each week clinicians and research staff meet to discuss the research projects that are currently being conducted and open to enrollment. Using this information, clinicians approach their patients they deem to be appropriate for research and that meet inclusion criteria. If a patient expresses interest in participating in research, the clinician completes a Clinician Referral Form and refers the patient to the appropriate research assistant for additional information regarding the study. A member of the research team will meet with the subject and explain the study protocol, including a review of risks and potential benefits.

Patients who express interest after this first meeting will be evaluated for competency to provide informed consent by a physician who is not a member of the research team. Competence to provide consent is assessed by a research psychiatrist using the Assessment of Capacity to Participate in Clinical Research form. Patients who are judged to be competent will then be asked to meet with the principal investigator who will review the study protocol and consent form with the patient and obtain informed consent. A copy of the study consent form will be provided to the patient at this time.

In addition, the prospective subject must ultimately score a 100% correct score on a True/False quiz about informed consent and the study they are interested in participating in.

Potential Risks:

Ziprasidone did not produce any serious adverse effects in animal and human safety studies. No consistent abnormality of vital signs, laboratory, or EEG has emerged. Prolongation of the QTC on EKG has been observed with ziprasidone treatment. In clinical trials, no side effects occurred at rates greater than 2x placebo. Nausea, vomiting, anxiety, headache, dyspepsia, somnolence, orthostatic hypotension, tachycardia, insomnia, akathisia, and EPS may be potential side effects.

Benefits:

It is not known if ziprasidone added to clozapine or olanzapine will help a subject's mood, motivation, hallucinations, and unusual experiences. Other patients may benefit if this study finds that ziprasidone added to clozapine or olanzapine is useful for treating symptoms of schizophrenia.

Protection of Human Subjects:

Principal members of our research team have all completed certification for protection of human subjects in clinical trials. The clinical protocol will be submitted for approval by the institutional review boards of the Massachusetts Department of Mental Health. Potential subjects will be referred by their clinicians. Clinicians will be asked to sign a statement that verifies that the patient is interested in participating, understands that participation is voluntary, and understands that declining participation will not affect treatment at the facility. A member of the research team will meet with the patient and explain the study protocol, including a review of risks and potential benefits. A copy of the study consent form will be provided to the patient at that time to share with family members or residential staff. Patients who continue to express interest after this first meeting will be evaluated by a physician for capacity to provide informed consent. Patients who are judged to be competent will then be asked to meet with the principal investigator or co-investigator who will review the study protocol and consent form with the patient and obtain informed consent.

Each subject that enrolls in the study is asked to sign an authorization to release information to their clinician. Upon consent, a letter is sent to the clinician with notification of study enrollment, the duration of the study and the dose and duration of any study medications.

All laboratory work and physical assessments performed during the study are either conducted or reviewed by a research physician. Side effects and vital signs are monitored routinely by the research assistants. Should any abnormal lab values or adverse events occur during the course of the subject's participation, the research physician would be notified immediately of these values and consulted on how to proceed with patient care. Furthermore, the subject's clinician would also be informed of the results.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia, any subtype or schizoaffective disorder
* Ages 18-65 years
* Capable of providing informed consent
* Antipsychotic Agents -associated diabetes mellitus, impaired fasting glucose or insulin resistance
* Stable dose of clozapine or olanzapine for at least 1 month
* Optimal dose of clozapine or olanzapine, or a maximal dose if limited by significant side effects

Exclusion Criteria:

* Serious medical or neurological illness (unstable cardiac disease including recent myocardial infarction or heart failure, seizure disorder, malignancy, liver or renal impairment, etc.)
* Current substance abuse
* Pregnancy, nursing, or unwilling to use appropriate birth control measures during participation if female and fertile
* History of serious blood dyscrasia requiring discontinuation of clozapine
* Serious suicidal or homicidal risk within the past six months
* History of diabetes mellitus prior to treatment with clozapine or olanzapine
* H/o prolongation of QTc interval (>450) on EKG or clinically significant EKG abnormalities.
* Treatment with medications that significantly prolong QTc interval such as dofetilde, sotalol, quinidine, class Ia and III antiarrhythmics, mesoridazine, thioridazine, chlorpromazine, droperidol, pimozide, sparfloxacin, gatifloxacin, moxifloxacine, halofantrine, mefloquine, pentamidine, arsenic trioxide, levomethadyul acetate, dolasetron myselate, probucol, or tacrolimus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-01; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Henderson, MD, Principal Investigator — North Suffolk Mental Health Association
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States

REFERENCES:
- [Background] Alao AO, Malhotra K, Dewan MJ. Comparing the side effect profile of the atypical antipsychotics. West Afr J Med. 2002 Oct-Dec;21(4):313-5. doi: 10.4314/wajm.v21i4.28008. PMID 12665274
- [Background] Allison DB, Mentore JL, Heo M, Chandler LP, Cappelleri JC, Infante MC, Weiden PJ. Antipsychotic-induced weight gain: a comprehensive research synthesis. Am J Psychiatry. 1999 Nov;156(11):1686-96. doi: 10.1176/ajp.156.11.1686. PMID 10553730
- [Background] Ananth J, Venkatesh R, Burgoyne K, Gunatilake S. Atypical antipsychotic drug use and diabetes. Psychother Psychosom. 2002 Sep-Oct;71(5):244-54. doi: 10.1159/000064807. PMID 12207104
- [Background] Baptista T, Kin NM, Beaulieu S, de Baptista EA. Obesity and related metabolic abnormalities during antipsychotic drug administration: mechanisms, management and research perspectives. Pharmacopsychiatry. 2002 Nov;35(6):205-19. doi: 10.1055/s-2002-36391. PMID 12518268
- [Background] Caro JJ, Ward A, Levinton C, Robinson K. The risk of diabetes during olanzapine use compared with risperidone use: a retrospective database analysis. J Clin Psychiatry. 2002 Dec;63(12):1135-9. doi: 10.4088/jcp.v63n1208. PMID 12523873
- [Background] Cohen S, Fitzgerald B, Okos A, Khan S, Khan A. Weight, lipids, glucose, and behavioral measures with ziprasidone treatment in a population with mental retardation. J Clin Psychiatry. 2003 Jan;64(1):60-2. doi: 10.4088/jcp.v64n0112. PMID 12590625
- [Background] Colli A, Cocciolo M, Francobandiera F, Rogantin F, Cattalini N. Diabetic ketoacidosis associated with clozapine treatment. Diabetes Care. 1999 Jan;22(1):176-7. doi: 10.2337/diacare.22.1.176a. No abstract available. PMID 10333925
- [Background] Daniel DG, Copeland LF. Ziprasidone: comprehensive overview and clinical use of a novel antipsychotic. Expert Opin Investig Drugs. 2000 Apr;9(4):819-28. doi: 10.1517/13543784.9.4.819. PMID 11060712
- [Background] Gianfrancesco FD, Grogg AL, Mahmoud RA, Wang RH, Nasrallah HA. Differential effects of risperidone, olanzapine, clozapine, and conventional antipsychotics on type 2 diabetes: findings from a large health plan database. J Clin Psychiatry. 2002 Oct;63(10):920-30. doi: 10.4088/jcp.v63n1010. PMID 12416602
- [Background] Goodnick PJ. Ziprasidone: profile on safety. Expert Opin Pharmacother. 2001 Oct;2(10):1655-62. doi: 10.1517/14656566.2.10.1655. PMID 11825308
- [Background] Green MF. What are the functional consequences of neurocognitive deficits in schizophrenia? Am J Psychiatry. 1996 Mar;153(3):321-30. doi: 10.1176/ajp.153.3.321. PMID 8610818
- [Background] Hagg S, Joelsson L, Mjorndal T, Spigset O, Oja G, Dahlqvist R. Prevalence of diabetes and impaired glucose tolerance in patients treated with clozapine compared with patients treated with conventional depot neuroleptic medications. J Clin Psychiatry. 1998 Jun;59(6):294-9. doi: 10.4088/jcp.v59n0604. PMID 9671341
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Henderson DC, Goff DC. Risperidone as an adjunct to clozapine therapy in chronic schizophrenics. J Clin Psychiatry. 1996 Sep;57(9):395-7. PMID 9746446
- [Background] Henderson DC, Cagliero E, Gray C, Nasrallah RA, Hayden DL, Schoenfeld DA, Goff DC. Clozapine, diabetes mellitus, weight gain, and lipid abnormalities: A five-year naturalistic study. Am J Psychiatry. 2000 Jun;157(6):975-81. doi: 10.1176/appi.ajp.157.6.975. PMID 10831479
- [Background] Kato MM, Goodnick PJ. Antipsychotic medication: effects on regulation of glucose and lipids. Expert Opin Pharmacother. 2001 Oct;2(10):1571-82. doi: 10.1517/14656566.2.10.1571. PMID 11825300
- [Background] Kay SR, Opler LA, Lindenmayer JP. Reliability and validity of the positive and negative syndrome scale for schizophrenics. Psychiatry Res. 1988 Jan;23(1):99-110. doi: 10.1016/0165-1781(88)90038-8. PMID 3363019
- [Background] Koller E, Schneider B, Bennett K, Dubitsky G. Clozapine-associated diabetes. Am J Med. 2001 Dec 15;111(9):716-23. doi: 10.1016/s0002-9343(01)01000-2. PMID 11747852
- [Background] Koller EA, Doraiswamy PM. Olanzapine-associated diabetes mellitus. Pharmacotherapy. 2002 Jul;22(7):841-52. doi: 10.1592/phco.22.11.841.33629. PMID 12126218
- [Background] Levine J, Schooler NR. SAFTEE: a technique for the systematic assessment of side effects in clinical trials. Psychopharmacol Bull. 1986;22(2):343-81. No abstract available. PMID 3774930
- [Background] Melkersson KI, Hulting AL, Brismar KE. Elevated levels of insulin, leptin, and blood lipids in olanzapine-treated patients with schizophrenia or related psychoses. J Clin Psychiatry. 2000 Oct;61(10):742-9. doi: 10.4088/jcp.v61n1006. PMID 11078035
- [Background] Newcomer JW, Haupt DW, Fucetola R, Melson AK, Schweiger JA, Cooper BP, Selke G. Abnormalities in glucose regulation during antipsychotic treatment of schizophrenia. Arch Gen Psychiatry. 2002 Apr;59(4):337-45. doi: 10.1001/archpsyc.59.4.337. PMID 11926934
- [Background] Nuechterlein KH, Dawson ME, Gitlin M, Ventura J, Goldstein MJ, Snyder KS, Yee CM, Mintz J. Developmental Processes in Schizophrenic Disorders: longitudinal studies of vulnerability and stress. Schizophr Bull. 1992;18(3):387-425. doi: 10.1093/schbul/18.3.387. PMID 1411329
- [Background] Opp D, Hildebrandt C. Olanzapine-associated type 2 diabetes mellitus. Schizophr Res. 2002 Jul 1;56(1-2):195-6. doi: 10.1016/s0920-9964(01)00226-2. No abstract available. PMID 12084434
- [Background] Pi-Sunyer FX. Medical hazards of obesity. Ann Intern Med. 1993 Oct 1;119(7 Pt 2):655-60. doi: 10.7326/0003-4819-119-7_part_2-199310011-00006. PMID 8363192
- [Background] Seaburg HL, McLendon BM, Doraiswamy PM. Olanzapine-associated severe hyperglycemia, ketonuria, and acidosis: case report and review of literature. Pharmacotherapy. 2001 Nov;21(11):1448-54. doi: 10.1592/phco.21.17.1448.34421. PMID 11714220
- [Background] Spivak B, Alamy SS, Jarskog LF, Sheitman BB, Lieberman JA. Ziprasidone alternative for olanzapine-induced hyperglycemia. Am J Psychiatry. 2002 Sep;159(9):1606. doi: 10.1176/appi.ajp.159.9.1606. No abstract available. PMID 12202289
- [Background] Taylor D. Ziprasidone in the management of schizophrenia : the QT interval issue in context. CNS Drugs. 2003;17(6):423-30. doi: 10.2165/00023210-200317060-00004. PMID 12697001
- [Background] Wetterling T. Bodyweight gain with atypical antipsychotics. A comparative review. Drug Saf. 2001 Jan;24(1):59-73. doi: 10.2165/00002018-200124010-00005. PMID 11219487
- [Background] Wilson DR, D'Souza L, Sarkar N, Newton M, Hammond C. New-onset diabetes and ketoacidosis with atypical antipsychotics. Schizophr Res. 2003 Jan 1;59(1):1-6. doi: 10.1016/s0920-9964(01)00331-0. PMID 12413635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will include 40 outpatients with schizophrenia or schizoaffective disorder treated with clozapine or olanzapine for at least one year. Twenty clozapine-treated subjects and twenty olanzapine-treated subjects with type 2 diabetes mellitus, impaired fasting glucose or insulin resistance will be recruited.
Pre-assignment Details: 24 subjects consented for the study. Two subjects consented but were lost to follow-up, and one subject withdrew consent after receiving one dose of ziprasidone.
Groups:
- Open-label Ziprasidone: All subjects will be treated with open label ziprasidone 40 mg 2x/day for the first 2 weeks. After 2 weeks the study drug may be increased up to ziprasidone 80 mg 2x/day. The subject's clozapine or olanzapine dose will be unchanged during the trial.
Period: Overall Study
Arm/Group | Open-label Ziprasidone
Started | 24
Completed | 21
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Ziprasidone
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (8)
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fasting Glucose
Description: Subjects on clozapine with adjunctive ziprasidone were compared to subjects on olanzapine with adjunctive ziprasidone on change in fasting glucose levels from baseline to study endpoint (week 6 - baseline)
Time Frame: baseline, week 6
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Clozapine Treatment With Adjunctive Ziprasidone: All subjects will be treated with open label ziprasidone 40 mg 2x/day for the first 2 weeks. After 2 weeks the study drug may be increased up to ziprasidone 80 mg 2x/day. The subject's clozapine dosage will be unchanged during the trial.
- Olanzapine Treatment With Adjunctive Ziprasidone: All subjects will be treated with open label ziprasidone 40 mg 2x/day for the first 2 weeks. After 2 weeks the study drug may be increased up to ziprasidone 80 mg 2x/day. The subject's olanzapine dosage will be unchanged during the trial.
Arm/Group | Clozapine Treatment With Adjunctive Ziprasidone | Olanzapine Treatment With Adjunctive Ziprasidone
Number analyzed (Participants) | 11 | 10
mg/dL | 5 (3) | -4.5 (9.1)
Statistical Analysis 1: Comparison: Clozapine Treatment With Adjunctive Ziprasidone; Test type: Superiority or Other; p = 0.956, t-test, 2 sided

2. Primary Outcome: Change From Baseline on Fasting Insulin
Description: Subjects on clozapine with adjunctive ziprasidone were compared to subjects on olanzapine with adjunctive ziprasidone on change in fasting insulin levels from baseline to study endpoint (week 6 - baseline)
Time Frame: baseline, week 6
Measure: Mean (Standard Deviation); unit: microIU/L
Groups:
- Clozapine Treatment With Adjunctive Ziprasidone; Olanzapine Treatment With Adjunctive Ziprasidone: All subjects will be treated with open label ziprasidone 40 mg 2x/day for the first 2 weeks. After 2 weeks the study drug may be increased up to ziprasidone 80 mg 2x/day. The subject's clozapine dose will be unchanged during the trial.
Arm/Group | Clozapine Treatment With Adjunctive Ziprasidone | Olanzapine Treatment With Adjunctive Ziprasidone
Number analyzed (Participants) | 11 | 10
microIU/L | 1 (4.5) | -0.9 (1.4)
Statistical Analysis 1: Comparison: Clozapine Treatment With Adjunctive Ziprasidone; Test type: Superiority or Other; p = 0.988, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Open-label Ziprasidone
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Ziprasidone (N=24)
difficulty breathing (Cardiac disorders) | 1 (1) — Subject brought himself to the MGH Emergency Room, complaining of weakness in the chest and trouble breathing. Assessed vital signs, EKG, and was given an IV solution. When vitals returned to normal, discharged with proscribed rest.
dizziness (General disorders) | 1 (1) — Subject went to Whidden Hospital and had blood work, EKG, EEG and MRI performed and all results were negative. Over the past 2 years she had experienced this symptom before. Discharged after 5 days with symptom recovered and no additional treatment.

LIMITATIONS AND CAVEATS:
The sample size in this study may not have been adequate to demonstrate the effectiveness of ziprasidone as an adjuvant therapy. The receptor-binding profile of ziprasidone may not significantly counteract the mechanisms of metabolic disturbances.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes